CLINICAL TRIAL: NCT02335775
Title: A Prospective Study of the Impact of Surgical and Pathologic Tissue Sampling Methods on Lymph Node Counts and Detection of Lymph Node Metastasis in Endometrial Cancer Staging
Brief Title: Lymph Node Counts in Endometrial Cancer Staging
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008993
Record Dates: First submitted 2014-12-15; First posted 2015-01-12 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purposes of this study are to determine whether total lymph node count or the percentage of identified nodes with metastatic disease are influenced by (1) the method of categorizing tissue specimens or (2) the techniques of pathologic processing following lymphadenectomy.

Patients with newly diagnosed endometrial carcinoma of high risk histologic type or uterine carcinosarcoma whose risk of LN metastasis exceeds 15% will be enrolled on this study. Patients will undergo staging to include hysterectomy and selective lymphadenectomy as per the clinical judgment of the primary Gynecologic Oncologist. Type of hysterectomy and the extent and distribution of lymphadenectomy is at the discretion of the surgeon. All patients will be scheduled for surgical staging. Each subject will have lymph nodes harvested on one side divided into specific basins, and on the contralateral side classified only as "pelvic" or "aortic". Surgical node specimens in the operating room will be labeled by (1) specific nodal basins on the randomly determined side as "external iliac", "obturator", "common iliac", "aortic", or "high aortic" and by (2) "pelvic" versus "aortic" (common iliac nodes will be considered as part of the "pelvic" specimen) on the contralateral side.

ELIGIBILITY:
Inclusion Criteria:

* Uterine cancer with one of the following pathologies: serous, clear cell, sarcoma or grade 3 differentiation
* surgical candidate

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Woman over the age of 18 diagnosed with grade 3, clear cell, serous or sarcoma types of endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Total gross node identification | 0-14 days post op
Percentage of lymph nodes showing metastatic cancer (%NM) | 0-14 days post op

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States